CLINICAL TRIAL: NCT05718739
Title: Assessing and Understanding Freezing of Gait At-home Environment: FOG@Home
Brief Title: Assessing and Understanding Freezing of Gait at Home: FOG@Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TASMC-23-RE-0072-CTIL
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Accelerometer; Video; Freezing of gait; Parkinson's disease; Detection and Prediction of FOG
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOG@Home (Experimental): Patients with Parkinson's disease who agreed to be monitored using cameras and acceleration measurements during daily life.
  Interventions: Device: AX6 6-axis logging accelerometer

INTERVENTIONS:
Device: AX6 6-axis logging accelerometer — The device is collecting longitudinal movement data.
  Other Names: AX6

SUMMARY:
Freezing of gait, (FOG) is an unpredictable, abrupt, short phenomenon that severely affects Parkinson's disease (PD) patients' gait and quality of life. The common measure tools are self-questioners that present the subjective feelings and the FOG provoking tests that used in clinic for evoking FOG and getting the estimated duration and the phenotype of the expressed phenomenon. The objective of this study is to investigate the FOG phenomenon using video cameras at patients' home with combination of wearable-axivity sensors and smart soles with a goal of objective assessment and quantification of freezing of gait severity in unsupervised daily-living environment of the PD patients.

DETAILED DESCRIPTION:
30 PD subjects, referred by the Movement Disorders Centre would be enrolled in the study according to eligibility criteria. By prior arrangement, the researchers will arrive to the participant's home. After explanation and consent process, the participant would sign the consent form. At that point, the patient would be assessed, before the execution of the experimental protocol. Hoehn and Yahr staging (H&Y), Unified Parkinson's Disease Rating Scale (UPDRS) and common cognitive tests would be applied. Then, the participant would be ask to put the motion sensors (accelerometers) and place the cameras in strategic places in the house, where he expect to see most freezing of gait events while walking around the house (no bedrooms and bathrooms). After activating the systems, the researchers would go, leaving the video system and the sensors for 7 days (depending on the amount of received data) in the patient house.

ELIGIBILITY:
Inclusion criteria:

Clinical diagnosis of Parkinson's disease (PD) according to the UK PD Society Brain Bank criteria; Modified Hoehn & Yahr Stage I to IV in the ON-state; Ability to walk 5 minutes while unassisted by another person; Mini-Mental State Examination (MMSE) score of >= 21 or > 16 on the 26-item MMSE screening; Self-reported freezing of gait (FOG) severity of at least 1 FOG episode per day, based on Characterizing of Freezing of Gait Questionnaire, irrespective of FOG occurring ON- or OFF-medication.

Exclusion criteria:

Acute musculoskeletal or other neurological or cardiovascular conditions affecting gait or any other medical condition which, in the opinion of the investigator, may prevent completing the protocol; The occurrence of any of the following within 3 months prior to informed consent: orthopedic surgery of the lower extremity, myocardial infarction, hospitalization for unstable angina, coronary artery bypass graft, percutaneous coronary intervention, implantation of a cardiac resynchronization therapy device, implantation of deep brain stimulation; Substance abuse, major depressive disorder or clinical apathy that affects daily walking activity or may interfere with the patient's compliance; Inability to walk without a rollator indoors; Absence of clinically observed FOG during the FOG-provoking assessment.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent with FOG (% FOG) during the monitoring period | immediate post monitoring
  The percentage of time spent with FOG (%FOG) can be obtained as an outcome from standardized gait assessments that are video-taped and scored offline for FOG episodes by a trained expert. Freezing includes episodes of akinetic FOG, trembling FOG and festination.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Alcalay, MD, Principal Investigator — Director of the Center for Movement Disorders, Neurological Department, Tel Aviv Sourasky Medical Center - Ichilov Hospital, Israel
Locations (1):
- Movement disorders unit, the Department of Neurology, Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giladi N, Nieuwboer A. Understanding and treating freezing of gait in parkinsonism, proposed working definition, and setting the stage. Mov Disord. 2008;23 Suppl 2:S423-5. doi: 10.1002/mds.21927. No abstract available. PMID 18668629
- [Result] Pardoel S, Kofman J, Nantel J, Lemaire ED. Wearable-Sensor-based Detection and Prediction of Freezing of Gait in Parkinson's Disease: A Review. Sensors (Basel). 2019 Nov 24;19(23):5141. doi: 10.3390/s19235141. PMID 31771246
- [Result] Gilat M. How to Annotate Freezing of Gait from Video: A Standardized Method Using Open-Source Software. J Parkinsons Dis. 2019;9(4):821-824. doi: 10.3233/JPD-191700. PMID 31524181
- [Result] Zoetewei D, Herman T, Brozgol M, Ginis P, Thumm PC, Ceulemans E, Decaluwe E, Palmerini L, Ferrari A, Nieuwboer A, Hausdorff JM. Protocol for the DeFOG trial: A randomized controlled trial on the effects of smartphone-based, on-demand cueing for freezing of gait in Parkinson's disease. Contemp Clin Trials Commun. 2021 Jun 29;24:100817. doi: 10.1016/j.conctc.2021.100817. eCollection 2021 Dec. PMID 34816053